CLINICAL TRIAL: NCT00055367
Title: A Phase II, International, Multicenter, Open Label Study of the Safety, Tolerability and Effectiveness of Three Intravenous Infusions of Antegren (Natalizumab) in Adolescents With Moderately to Severely Active Crohn's Disease
Brief Title: Safety, Tolerability and Effectiveness of Natalizumab in Adolescents With Active Crohn's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biogen (Industry)
Collaborators: Elan Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CD305
Record Dates: First submitted 2003-02-26; First posted 2003-02-28 (Estimated); Last update posted 2016-06-16 (Estimated); Status verified 2012-03

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — Natalizumab

INTERVENTIONS:
Drug: natalizumab

SUMMARY:
The purpose of this study is to determine the safety and tolerability of natalizumab in adolescents (ages 12-17) diagnosed with moderately to severely active Crohn's disease (CD). It is thought that natalizumab may stop the movement of certain cells, known as white blood cells, into bowel tissue. These cells are thought to cause damage in the bowel leading to the symptoms of Crohn's disease.

Patients who complete this study may be eligible for long-term natalizumab therapy via extension protocol ELN100226-352.

ELIGIBILITY:
Male and female patients, 12-17 years of age, who have at least a six-month history of Crohn's disease and who are currently experiencing moderately to severely active Crohn's disease. Females must not be breastfeeding or pregnant, and must not become pregnant during the study.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30
Dates: Start 2002-04; Primary Completion 2004-05 (Actual); Study Completion 2004-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (13):
- United States (11):
  - Cedars-Sinai IBD Center, Los Angeles, California
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Miami Research Associates, Miami, Florida
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Mass General Hospital for Children, Pediatric GI & Nutrition, Boston, Massachusetts
  - The Children's Hospital, Boston, Massachusetts
  - University of Rochester, Rochester, New York
  - Carolina Digestive Health Associates, Charlotte, North Carolina
  - Hershey Medical Center, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- United Kingdom (2):
  - Royal Hospital for Sick Children, Edinburgh
  - Royal Free Medical School, London